CLINICAL TRIAL: NCT06377631
Title: Effect of a Multi-ingredient of L-Histidine, L-Serine, L-Carnosine and N-Acetylcysteine on Visceral Adiposity and Non-alcoholic Fatty Liver Disease in Postmenopausal Women With Abdominal Obesity
Brief Title: Effect of Multi-ingredient on Visceral Adiposity & Non-alcoholic Fatty Liver Disease in Postmenopausal Women With Abdominal Obesity
Acronym: FATHIS+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Eurecat (Other)
Collaborators: Centre de Diagnosi per la Imatge (Unknown); Instituto de Investigación Biomédica de Girona (IDIBGI) (Unknown); Laboratorio de Referencia de Cataluña (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FATHIS+
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Visceral Obesity; Non-alcoholic Fatty Liver; Postmenopausal
Keywords: Nutraceuticals; Metabolic risk; Visceral obesity; NAFLD; Hepatic steatosis; Lipid metabolism; Cardiovascular risk; Postmenopause; Histidine
MeSH Terms: conditions — Obesity, Abdominal; Non-alcoholic Fatty Liver Disease; Fatty Liver | interventions — Serine; Carnosine; Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multi-ingredient of L-histidine, L-serine, L-carnosine and N-Acetylcysteine (Experimental): Participants will daily consume the multi-ingredient (L-Histidine, L-Serine, L-Carnosine and N-Acetylcysteine) for 12 weeks.
  Interventions: Dietary Supplement: Multi-ingredient of L-histidine, L-serine, L-carnosine and N-Acetylcysteine
- Placebo (Placebo Comparator): Participants will daily consume the placebo (maltodextrin) for 12 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Multi-ingredient of L-histidine, L-serine, L-carnosine and N-Acetylcysteine — The product will be presented in powder format in a single container and with a measuring spoon of the daily dose.
  Arms: Multi-ingredient of L-histidine, L-serine, L-carnosine and N-Acetylcysteine
Dietary Supplement: Placebo — The product will be presented in powder format in a single container and with a measuring spoon of the daily dose.
  Arms: Placebo

SUMMARY:
This study aims to evaluate the effect of daily intake of a specific combination of different natural histidine-related amino acids in combination with dietary recommendations, in the reduction of visceral fat, as well as their associated comorbidities, in postmenopausal women with abdominal obesity.

DETAILED DESCRIPTION:
In postmenopausal women, the risk of non-alcoholic fatty liver disease (NAFLD) increases due to hormonal changes and metabolic shifts. Menopause leads to a decline in estrogen levels, affecting lipid metabolism and promoting abdominal and visceral fat accumulation. This visceral adiposity poses a significant risk factor for insulin resistance, type 2 diabetes, dyslipidemia, cardiovascular diseases, and NAFLD. While the prevalence of NAFLD is initially higher in men, it becomes comparable or even higher in postmenopausal women due to these metabolic changes.

Studies suggest that estrogen deficiency post-menopause contributes to the development of NAFLD in women. Lower serum estrogen levels are associated with a higher likelihood of NAFLD development, indicating the potential role of hormone replacement therapy (HRT) in mitigating NAFLD risk in postmenopausal women. However, the use of HRT must be carefully evaluated due to potential adverse effects on cardiovascular health.

Thus, novel, effective and safety therapeutic strategies for managing metabolic disorders in postmenopausal women are highly desirable.

The main objective of this study is to evaluate the effect of daily intake of a specific combination of different natural histidine-related amino acids in combination with dietary recommendations, in the reduction of visceral fat in postmenopausal women with abdominal obesity.

The secondary objectives of this study are to evaluate the effect of daily intake of the multi-ingredient aforementioned in liver function markers, anthropometric parameters, blood pressure and heart rate, markers of lipid metabolism, markers of glucidic metabolism, inflammatory markers, histidine serum levels, sexual hormones, the temperature of supraclavicular brown adipose tissue, changes in the intestinal microbiota, changes in the expression of lipid metabolism-related genes and symptoms associated with postmenopause.

A randomized, parallel, placebo-controlled, single-center, triple-blind clinical trial with a 1:1:1 ratio between interventions with 50 participants will be conducted.

During the study there will be 4 visits: a preselection visit (V0; day -7) and 3 study visits during the consumption of the treatments, which will take place on the first day of the study (V1; day 1 +/- 3 days; week 1), at 6 weeks of treatment (V2; day 43 +/- 3 day; week 6) and at 12 weeks of treatment (V3; day 85 +/- 3 days; week 12).

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women aged 50 to 65 years.
* BMI ≥27.5 kg/m^2 and ≤32.5 kg/m^2.
* Waist circumference ≥88 cm.
* No hormone replacement therapy.
* Read, write and speak Catalan or Spanish.
* Sign the informed consent.

Exclusion Criteria:

* Present values of body mass index < 27.5 kg/m^2 or > 32.5 kg/m^2
* Present values of waist circumference > 115 cm.
* Present diabetes.
* Present dyslipidemia.
* Present anemia.
* Taking supplements, multivitamin supplements or phytotherapeutic products that interfere with the treatment under study.
* Consume 2 or more Standard Beverage Units (SBU) daily or 17 SBU weekly.
* Be a smoker.
* Present any diagnosed liver disease other than NAFLD.
* Have lost more than 3 kg of weight in the last 3 months.
* Present food intolerances and/or allergies related to the study products, such as hypersensitivity to maltodextrin or N-Acetylcysteine.
* Presenting any chronic or autoimmune disease in clinical manifestation such as hepatitis, hyper or hypothyroidism or metabolic diseases.
* Follow a pharmacological treatment with immunosuppressants, cytotoxic agents, corticosteroids or other drugs that could cause hepatic steatosis or alter the measurements in the liver.
* Being participating or having participated in a clinical trial or nutritional intervention study in the last 30 days before inclusion in the study.
* Follow a hypocaloric diet and/or pharmacological treatment for weight loss.
* Suffering from eating behavior disorders or psychiatric disorders.
* Being unable to follow study guidelines.

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-06-07 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2025-04-08 (Actual)

PRIMARY OUTCOMES:
Change in Visceral Adiposity | Change from Baseline Visceral Adiposity at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Visceral fat content measured using a dual energy x-ray absorptiometry (DXA) scanner

SECONDARY OUTCOMES:
Height (cm) | At baseline
  Height measured with standardized method
Age | At day -7 (pre-selection visit)
  The age of the volunteers will be recorded in the case report form.
Ethnicity | At day -7 (pre-selection visit)
  The ethnicity of the volunteers will be recorded in the case report form.
Change in Body Weight (kg) | Change from Baseline Weight at 6 and 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Weight measured with standardized method
Change in Body Mass Index (BMI) (Kg/m^2) | Change from Baseline Body Mass Index at 6 and 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Weight and height will be combined to report BMI in kg/m^2
Change in Neck circumference (cm) | Change from Baseline Neck circumference at 6 and 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Neck circumference using a measuring tape
Change in Arm circumference (cm) | Change from Baseline Arm circumference at 6 and 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Arm circumference using a measuring tape
Change in Waist circumference (cm) | Change from Baseline Waist circumference at 6 and 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Waist circumference using a measuring tape
Change in Hip circumference (cm) | Change from Baseline hip circumference at 6 and 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Hip circumference using a measuring tape
Change in Conicity Index | Change from Baseline Conicity Index at 6 and 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Weight, height and waist circumference will be combined to report Conicity index.
Change in Waist-to-Hip ratio | Change from Baseline Waist-to-Hip ratio at 6 and 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Waist and Hip circumference will be combined to report Waist-to-Hip ratio
Change in Lipid Accumulation Product (LAP) | Change from Baseline Lipid Accumulation Product ratio at 6 and 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Waist circumference and fasting plasma Triglycerides will be combined to report Lipid Accumulation Product
Change in Systolic Blood Pressure (mm Hg) | Change from Baseline Systolic Blood Pressure at 6 and 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Systolic blood pressure will be measured using an automatic sphygmomanometer
Change in Diastolic Blood Pressure (mm Hg) | Change from Baseline Systolic Blood Pressure at 6 and 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Diastolic blood pressure will be measured using an automatic sphygmomanometer
Change in heart rate (bpm) | Change from Baseline Heart rate at 6 and 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Heart rate will be measured using an automatic sphygmomanometer
Change in serum glucose levels (mg/dL) | Change from Baseline serum glucose levels at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Serum glucose levels will be determined by standardized spectrophotometry methods
Change in serum total cholesterol (mg/dL) | Change from Baseline serum total cholesterol at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Total cholesterol will be determined by standardized spectrophotometry methods
Change in serum high-density lipoprotein cholesterol (HDL-C,mg/dL) | Change from Baseline serum high-density lipoprotein cholesterol at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  High-density lipoprotein cholesterol will be determined by standardized spectrophotometry methods
Change in serum low-density lipoprotein cholesterol (LDL-C, mg/dL) | Change from Baseline serum low-density lipoprotein cholesterol at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Low-density lipoprotein cholesterol will be calculated using the Friedewald formula
Change in serum triglycerides (TG, mg/dL) | Change from Baseline serum triglycerides at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Triglycerides will be determined by standardized spectrophotometry methods
Change in serum alanine aminotransferase (ALT, U/L) | Change from Baseline serum alanine aminotransferase at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Alanine aminotransferase will be determined by standardized spectrophotometry methods
Change in serum aspartate aminotransferase (AST, U/L) | Change from Baseline serum aspartate aminotransferase at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Aspartate aminotransferase will be determined by standardized spectrophotometry methods
Change in serum gamma glutamyl transferase (GGT, U/L) | Change from Baseline serum gamma glutamyl transferase at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Gamma glutamyl transferase will be determined by standardized spectrophotometry methods
Change in serum insulin levels (mU/L) | Change from Baseline serum insulin levels at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Insulin levels will be measured by standardized chemiluminescence methods.
Change in serum leptin levels (pg/mL) | Change from Baseline serum leptin levels at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Leptin levels will be measured by standardized chemiluminescence methods
Change in serum adiponectin levels (ng/mL) | Change from Baseline serum adiponectin levels at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Adiponectin levels will be measured by standardized chemiluminescence methods
Change in Adiponectin/Leptin ratio (numerical ratio) | Change from Baseline Adiponectin/Leptin ratio at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Adiponectin and leptin will be combined to report adiponectin/leptin ratio
Change in serum Monocyte chemoattractant protein-1 (MCP-1) levels (pg/mL) | Change from Baseline serum MCP-1 levels at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  MCP-1 levels will be measured by standardized chemiluminescence methods
Change in plasma tumor necrosis factor alpha (TNF-alpha) levels (pg/mL) | Change from Baseline plasma TNF-alpha levels at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  TNF-alpha levels will be measured by standardized chemiluminescence methods
Change in plasma Interleukin 6 (IL-6) levels (pg/mL) | Change from Baseline plasma IL-6 levels at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  IL-6 levels will be measured by standardized chemiluminescence methods
Change in plasma Interleukin 10 (IL-10) levels (pg/mL) | Change from Baseline plasma IL-10 levels at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  IL-10 levels will be measured by standardized chemiluminescence methods
Change in plasma Intercellular Adhesion Molecule 1 (ICAM-1) levels (ng/mL) | Change from Baseline plasma ICAM-1 levels at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  ICAM-1 levels will be measured by standardized chemiluminescence methods
Change in plasma Cluster of Differentiation 14 (CD14) levels (pg/mL) | Change from Baseline plasma CD14 levels at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  CD14 levels will be measured by standardized chemiluminescence methods
Change in plasma oxidized low density lipoproteins (LDLox) levels (mU/L) | Change from Baseline plasma LDLox levels at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  LDLox levels will be measured by standardized chemiluminescence methods
Change in serum C-Reactive protein levels (mg/L) | Change from Baseline serum C-Reactive protein levels at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  C-Reactive protein levels will be determined by standardized spectrophotometry methods
Change in Histidine levels in blood (umol/L) | Change from Baseline Histidine levels at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Serum histidine levels will be determined by Liquid Chromatography coupled to tandem Mass Spectrometry
Change in Acylcarnitine levels in blood (umol/L) | Change from Baseline Acylcarnitine levels at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Serum Acylcarnitine levels will be determined by Liquid Chromatography coupled to tandem Mass Spectrometry
Change in 17-beta-estradiol (E2) levels in blood (pg/mL) | Change from Baseline 17-beta-estradiol (E2) levels at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Serum 17-beta-estradiol (E2) levels will be determined by standardized chemiluminescence methods
Change in Follicle-stimulating hormone (FSH) levels in blood (mU/mL) | Change from Baseline FSH levels at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Follicle-stimulating hormone (FSH) levels will be determined by standardized chemiluminescence methods
Change in Homeostatic Model Assessment from Insulin Resistance Index (HOMA-IR) | Change from Baseline HOMA-IR at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  HOMA-IR will be calculated using serum glucose and insulin levels.
Change in Fatty Liver Index (FLI) | Change from Baseline FLI at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  FLI will be calculated using BMI, waist circumference, serum triglycerides and gamma glutamyl transferase levels
Change in Triglyceride glucose index (TyG) | Change from Baseline TyG at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  TyG will be calculated using serum glucose and triglycerides levels
Change in Plasma atherogenic index | Change from Baseline Plasma atherogenic index at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Plasma atherogenic index will be calculated as the logarithm of the TG to HDL-c ratio
Change in lipidomic profile | Change from Baseline Lipidomic profile at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Lipidomic analyses will be done by Liquid Chromatography coupled to tandem Mass Spectrometry
Change in intestinal microbiota composition | Change from Baseline intestinal microbiota composition at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Metagenomic analysis in fecal samples. The bacteria DNA will be extracted and massive sequenced by the Ion Torrent platform.
Change in the expression of lipid-metabolism genes in PBMC | Change from Baseline gene expression at 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Peripheral blood mononuclear cell (PBMC) will be isolated to obtain the RNA for gene expression analyses by Quantitative reverse transcription PCR (RT-qPCR)
Change in Dietary habits | Change from Baseline Dietary habits at 6 and 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Nutritional habits will be determined based on the results obtained from the 3-day dietary record
Change in Physical activity | Change from Baseline Physical activity at 6 and 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Physical activity will be evaluated through the International Physical Activity Questionnaire (IPAQ)-short for physical activity questionnaire. Scores will be reported in categories: LOW activity levels, MODERATE activity levels or HIGH activity levels with the latter indicating better outcomes.
Concomitant medication | At day -7 (pre-selection visit), day 1 (visit V1), day 43 (visit 2) and day 85 (visit 3)
  Concomitant medication consumed during the study will be recorded in the case report form.
Consumption of dietary supplements | At day -7 (pre-selection visit), day 1 (visit V1), day 43 (visit 2) and day 85 (visit 3)
  Dietary supplements consumed during the study will be recorded in the case report form.
Change in the Supraclavicular skin temperature | Change from Baseline Supraclavicular skin temperature at 6 and 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Supraclavicular skin temperature will be measured with the FLIR T530 thermal imaging camera
Change in postmenopausal symptoms | Change from Baseline postmenopausal symptoms at 6 and 12 weeks for each of the two treatments (multi-ingredient and placebo)
  Postmenopausal symptoms will be evaluated through the Menopause Rating Scale (MRS) questionnaire. The MRS comprises 11 items representing various symptoms or complaints. Each symptom can be rated from 0 (indicating no complaints) to 4 points (indicating severe symptoms), depending on the perceived severity reported by the women completing the scale. The total MRS score ranges from 0 (asymptomatic) to 44 (maximum complaint severity).
Adverse events | At 6 weeks (V2) and at 12 weeks (V3) for each of the two treatments (multi-ingredient and placebo)
  Possible adverse events derived from taking study's products will be recorded in the case report form

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Caimari, PhD, Principal Investigator — Fundació Eurecat
Locations (2):
- Spain (2):
  - Anna Crescenti, Reus, Catalonia. Spain
  - Fundació Eurecat, Reus, Tarragona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Technological Centre of Nutrition and Health. Eurecat_Reus. — http://eurecat.org